CLINICAL TRIAL: NCT04479527
Title: Evaluation Effectiveness and Safety of (cTACE or DEB-TACE + FOLFOX Regimen HAIC) Combined With Camrelizumab and Apatinib Mesylas in the Treatment of Advanced Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: Jiangsu Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Zhu Xu, Chief Physician, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20200705
Record Dates: First submitted 2020-07-13; First posted 2020-07-21 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2020-07

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — camrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- the group of HAIC combined with carilizumab and apatinib mesylate treatment (Experimental): cTACE or DEBTACE+FOLFOX scheme HAIC, arterial chemotherapy scheme: OXA 65-85mg/m2 arterial H0-4 pump, calcium folinate 200mg/ m2 intravenous pump H2-4, 5-FU 1g-1.5g/ m2 arterial H4-24 pump, once every 6-8 weeks, the interventional treatment times are determined by researchers according to the patient's condition, and two times are adjacent.
  Apatinib mesylate tablets, 250mg/ time, once a day. Take it about half an hour after a meal (the daily medication time should be as same as possible), and take it with warm boiled water.
  Karelizumab, 200mg, was given intravenously for 30 minutes (including the flushing time, the whole infusion time was not shorter than 20 minutes and not longer than 60 minutes), and the medication period was q3w(±3 days).
  Interventions: Drug: Camrelizumab

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab for injection is used to treat patients with relapsed or refractory classic Hodgkin lymphoma who have undergone at least second-line chemotherapy. Approved by the Drug Administration (NMPA) on March 4, 2020, for the treatment of patients with advanced hepatocellular carcinoma who have previously received sorafenib therapy and/or oxaliplatin-containing chemotherapy.Apatinib Mesylas is a small-molecule VEGFR tyrosine kinase inhibitor. It mainly treats malignant tumors by inhibiting VEGFR to play an anti-angiogenic effect. It has been approved by the China Food and Drug Administration (CFDA) in November 2014. It is used as a monotherapy for advanced gastric adenocarcinoma or gastric-esophageal junction adenocarcinoma that has progressed or relapsed after receiving two kinds of systemic chemotherapy. Apatinib Mesylas can effectively inhibit VEGFR2 at very low concentrations, and higher concentrations can also inhibit PDGFR, c-Kit and c-Src and other kinases.
  Other Names: Apatinib Mesylas

SUMMARY:
This study used (cTACE or DEB-TACE + FOLFOX scheme HAIC) combined with PD-1 antibody camrelizumab and apatinib mesylas in the treatment of patients with advanced liver cancer, to evaluate the effectiveness and safety of the combined treatment for clinical liver cancer treatment.It will provide new evidence-based medical evidence.This study is a prospective, open, single center, exploratory clinical study and the sample size is 56.Main research purpose:To evaluate the effectiveness of cTACE or DEB-TACE + FOLFOX regimen HAIC combined with camrelizumab and apatinib mesylas in the treatment of advanced hepatocellular carcinoma.Secondary research purpose:To evaluate the safety of cTACE or DEB-TACE + FOLFOX regimen HAIC combined with camrelizumab and apatinib mesylas in the treatment of advanced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75 years old, male or female;
2. Patients with primary hepatocellular carcinoma diagnosed by pathological or cytological examination;
3. Child-Pugh score: Grade A or better Grade B (≤7 points);
4. Surgical resection or local ablation is impossible. Patients with bclc stage b and c with ≥7 nodules or > 5 cm nodules;
5. PS score within one week before entering the group: 0-1;
6. There are measurable lesions that meet the mRECIST standard;
7. The main organs function normally, that is, they meet the following standards:

(1) routine blood examination:

1. HB≥90 g/L；
2. ANC≥1.5×109/L；
3. PLT≥100×109/L； (2) Biochemical examination:

a)ALB ≥29g/L； B)ALT and ast < 3 uln; c)TBIL ≤1.5ULN； D) creatinine ≤ 1.5 uln; 8. Women of childbearing age (generally 15-49 years old) must have a negative pregnancy test (serum or urine) within 14 days before entering the group, and voluntarily adopt appropriate methods of contraception during the observation period and within 8 weeks after the last administration of research drugs; For men, they should be sterilized by surgery or agree to use appropriate methods of contraception during the observation period and within 8 weeks after the last administration of study drugs.

Exclusion Criteria:

1. Patients with known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation or planned transplantation;
2. The previous use of immunosuppressive drugs within 14 days before the first use of Karelizumab, excluding nasal and inhaled corticosteroids or systemic steroid hormones with physiological dose (i.e. prednisolone or other corticosteroids with the same physiological dose);
3. It is known to be allergic to apatinib, kareli zumab or pharmaceutical excipients; Or severe allergic reaction to other monoclonal antibodies;
4. Vaccinate live attenuated vaccine within 4 weeks before the first administration or during the study period;
5. There are peripheral neuropathy of grade > 1;
6. There are any active autoimmune diseases or a history of autoimmune diseases;
7. Any other malignant tumor that has been diagnosed, except basal cell or squamous cell skin cancer or cervical carcinoma in situ that has been fully treated;
8. Human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS), active hepatitis B (HBV DNA ≥ 1000 IU/ml), hepatitis C (hepatitis C antibody is positive, and HCV-RNA is higher than the detection limit of analysis method) or combined with hepatitis B and hepatitis C co-infection;
9. Within 6 months before entering the study, the following conditions occurred: myocardial infarction, severe/unstable angina pectoris, NYHA 2 or above cardiac insufficiency, arrhythmia with poor control (including QTcF interval > 450 ms for men and > 470 ms for women, QTcF interval calculated by Fridericia formula), symptomatic congestive heart failure;
10. Hypertension, which cannot be well controlled by antihypertensive drug treatment (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥ 90 mmHg);
11. Abnormal coagulation function (INR>1.5 or APTT>1.5×ULN), bleeding tendency or being treated with thrombolytic therapy, anticoagulant therapy or antiplatelet therapy, etc.;
12. It is known that there are hereditary or acquired bleeding and thrombotic tendencies, such as hemophilia, coagulation dysfunction, thrombocytopenia, hypersplenism, etc.;
13. There is obvious cough blood within 2 months before entering the study, or the daily cough blood volume reaches half a teaspoon (2.5 ml) or more;
14. Patients with gastrointestinal bleeding risk, including the following:

(1) Active peptic ulcer lesions; (2) Those who have a history of black stool and hematemesis within 3 months; (3) For fecal occult blood (+) or (+/-), it needs to be reviewed within 1 week, and gastroscopy should be performed if it is still (+) or (+/-). If there is ulcer or hemorrhagic disease, and the attending doctor thinks there is potential bleeding risk; 15. Arterial/venous thrombosis events occurred within 6 months before entering the study, such as cerebrovascular accidents (including temporary ischemic attack, cerebral hemorrhage and cerebral infarction), deep venous thrombosis and pulmonary embolism, etc.; 16. Infections requiring drug intervention within 4 weeks before the first administration (such as intravenous drip of antibiotics, antifungal or antiviral drugs), or fever of unknown cause > 38.5°C； during screening/before the first administration; 17. Participated in any other drug clinical research within 4 weeks before the first administration; 18. It is known that there is a history of psychotropic drug abuse or drug abuse; There are other serious physical or mental diseases or abnormal laboratory examination, which may increase the risk of participating in the study, or interfere with the results of the study, and the researchers think that the patients are not suitable for participating in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | Up to 2 years.
  PFS refers to the length of time from the beginning of treatment to disease progression or death for any reason.

SECONDARY OUTCOMES:
ORR | Up to 2 years.
  The objective response rate (ORR) refers to the proportion of patients whose tumor volume has reduced to a predetermined value and can maintain the minimum time limit.
DCR | Up to 2 years.
  Disease control rate (DCR) refers to the proportion of patients whose tumors shrink or stabilize and remain for a certain period of time, including cases with complete response (CR), partial response (PR), and stable (SD).
OS | Up to 2 years.
  Overall survival (OS) refers to the time from enrollment to death due to any cause.
Incidence of AE and SAE | Up to 2 years.
  All adverse events in all subjects in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Xu Zhu, MD, Principal Investigator — Peking University Cancer Hospital & Institute; Xiaodong Wang, MD, Principal Investigator — Peking University Cancer Hospital & Institute